CLINICAL TRIAL: NCT07122388
Title: "Retrospective Study on the Evaluation of Sleep Habits, Sleep Macrostructure and Microstructure in Children and Adolescents With Autism Spectrum Disorder: Association With Behavioral Variables and Parental Stress"
Brief Title: "Sleep Patterns and EEG Structure in Youth With Autism: Links With Behavior and Parental Stress"
Status: Active, not recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Marco Carotenuto, Full Professor of Child Neuropsychiatry, University of Campania Luigi Vanvitelli
Other Study IDs: 217
Record Dates: First submitted 2025-07-30; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Sleep Disorder (Disorder); Autism Spectrum Disorder
Keywords: NREM sleep instability; CAP analysis; CBCL; ADOS-2; ADI-R; PSI-SF; Polysomnography
MeSH Terms: conditions — Sleep Wake Disorders; Autism Spectrum Disorder | interventions — Sleep; Polysomnography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autism spectrum disorder: Subjects with SRS-2 positive screening and confirmed by ADOS-2 evaluation
  Interventions: Diagnostic Test: Questionnaires about autism spectrum disorders and sleep and PSG.; Diagnostic Test: ADOS-2, ADI-R, SRS-2, PSG

INTERVENTIONS:
Diagnostic Test: Questionnaires about autism spectrum disorders and sleep and PSG. — Recruitment of subjects with autism spectrum disorder at all developmental ages and of all severity levels.
Diagnostic Test: ADOS-2, ADI-R, SRS-2, PSG — Recruitment of subjects with autism spectrum disorder at all developmental ages and all severity levels.

SUMMARY:
This retrospective observational study is designed to investigate sleep patterns, as well as both the macrostructure and microstructure of sleep, in a large cohort of children and adolescents diagnosed with Autism Spectrum Disorder (ASD). The study will utilize data derived from overnight polysomnographic recordings, providing objective and comprehensive measures of sleep architecture.

The sample consists of 187 patients, aged between 3 and 16 years, whose sleep data were collected over a ten-year period, from 2003 to 2013. In addition to polysomnographic parameters, the study will incorporate a wide range of behavioral and parental stress-related variables. These will be assessed using validated, standardized instruments, including the Sleep Disturbance Scale for Children (SDSC), Autism Diagnostic Interview-Revised (ADI-R), Autism Diagnostic Observation Schedule-2 (ADOS-2), Child Behavior Checklist (CBCL), and the Parenting Stress Index - Short Form (PSI-SF).

By integrating objective sleep data with behavioral and psychosocial measures, this study aims to provide a more nuanced understanding of the nature and extent of sleep disturbances in individuals with ASD. Particular attention will be paid to identifying potential correlations between specific sleep alterations (e.g., changes in sleep efficiency, REM latency, arousals, or cyclic alternating patterns) and behavioral symptoms or parental stress profiles.

Ultimately, the findings are expected to contribute to the development of more precise and individualized diagnostic frameworks, as well as inform evidence-based therapeutic strategies. These insights could be of considerable clinical relevance, given the high prevalence of sleep disorders in the ASD population and their significant impact on daytime functioning, emotional regulation, and family quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder
* Age: 3-18 years
* Sex: Both male and female
* Individuals with Autism Spectrum Disorder, including both verbal and non-verbal subjects
* Individuals with Autism Spectrum Disorder, with or without a comorbid genetic syndrome or other neurodevelopmental disorders

Exclusion Criteria:

* Neuropsychiatric disorders other than autism
* Epilepsy
* Age under 3 years or over 18 years
* Comorbidity with another severe psychiatric disorder (e.g., psychosis, schizophrenia)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adolescents with autism spectrum disorder
Sampling Method: Non-Probability Sample
Enrollment: 187 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
This retrospective observational study aims to evaluate sleep habits, as well as sleep macrostructure and microstructure, in a large cohort of children and adolescents with Autism Spectrum Disorder (ASD) through overnight polysomnographic assessment. | Baseline (single night recording)
  Assessment of sleep architecture parameters scored according to the American Academy of Sleep Medicine (AASM) pediatric criteria.
Total Sleep Time (TST) measured in minutes by overnight polysomnography | Baseline (single night recording)
  otal sleep time will be calculated from a single-night video-polysomnography recording, scored according to American Academy of Sleep Medicine (AASM) pediatric criteria.
Sleep Latency measured in minutes by overnight polysomnography | Baseline (single night recording)
  Sleep latency will be calculated as the time from lights-off to the first epoch of any sleep stage, scored according to AASM pediatric criteria.
Sleep Efficiency measured as a percentage by overnight polysomnography | Baseline (single night recording)
  Sleep efficiency will be calculated as the ratio of total sleep time to total time in bed, expressed as a percentage, scored according to AASM pediatric criteria.
Percentage of time spent in N1, N2, N3, and REM stages measured by overnight polysomnography | Baseline (single night recording)
  The proportion of total sleep time spent in each sleep stage will be calculated and expressed as a percentage, scored according to AASM pediatric criteria.
Duration of N1, N2, N3, and REM stages measured in minutes by overnight polysomnography. | Baseline (single night recording)
  The absolute duration of each sleep stage will be calculated in minutes, scored according to AASM pediatric criteria.

SECONDARY OUTCOMES:
Microstructural Sleep Parameters - Cyclic Alternating Pattern (CAP) Analysis from Overnight Polysomnography | Baseline (single night recording)
  Quantitative analysis of sleep microstructure, including CAP rate, phase A subtypes, and non-CAP periods, according to Terzano et al. methodology.
Sleep Habits - Sleep Disorders Scale for Children (SDSC) | Baseline
  Parent-completed 26-item questionnaire assessing six dimensions of sleep disturbances in children and adolescents over the previous 6 months.
Parental Stress - Parenting Stress Index Short Form (PIS-SF) | Baseline
  36-item questionnaire assessing parental distress, parent-child dysfunctional interaction, and perceptions of the child's temperament.
Social Impairment - Autism Diagnostic Interview-Revised (ADI-R) | Baseline
  Structured parent interview assessing qualitative abnormalities in reciprocal social interaction, communication, and restricted/repetitive behaviors.
Autism Severity - Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) | Baseline
  Standardized, semi-structured observational assessment used to classify autism severity levels (1, 2, or 3) according to DSM-5 criteria.
Behavioral Assessment - Child Behavior Checklist (CBCL; Age-Specific Parent-Report Forms) | Baseline
  Parent-report questionnaire assessing a wide range of emotional and behavioral problems in children aged 1-5 or 6-18 years.
Demographics - Age and Sex | Baseline
  Participant age (in years) and sex (male, female).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Napoli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marotta R, Risoleo MC, Messina G, Parisi L, Carotenuto M, Vetri L, Roccella M. The Neurochemistry of Autism. Brain Sci. 2020 Mar 13;10(3):163. doi: 10.3390/brainsci10030163. PMID 32182969
- [Background] Voci A, Mazzone L, De Stefano D, Valeriani M, Bruni O, Moavero R. Restless sleep disorder in a sample of children and adolescents with autism spectrum disorder: preliminary results from a case series. J Clin Sleep Med. 2024 Mar 1;20(3):427-432. doi: 10.5664/jcsm.10902. PMID 37909101
- [Background] Belli A, Breda M, Di Maggio C, Esposito D, Marcucci L, Bruni O. Children with neurodevelopmental disorders: how do they sleep? Curr Opin Psychiatry. 2022 Sep 1;35(5):345-351. doi: 10.1097/YCO.0000000000000790. Epub 2022 Feb 15. PMID 35165244
- [Background] Bernardi K, Prono F, Bruni G, Panerai S, Ferri R, Bruni O. Sleep disturbances in subjects with autism spectrum disorder: A parental perspective. Sleep Med. 2023 Oct;110:220-224. doi: 10.1016/j.sleep.2023.08.020. Epub 2023 Aug 23. PMID 37643569
- [Background] Bruni O, Breda M, Mammarella V, Mogavero MP, Ferri R. Sleep and circadian disturbances in children with neurodevelopmental disorders. Nat Rev Neurol. 2025 Feb;21(2):103-120. doi: 10.1038/s41582-024-01052-9. Epub 2025 Jan 8. PMID 39779841
- [Background] Scahill L, Johnson CR, Wenzell ML, Barto LM, Mulligan A, Williams AT, Johnson LM, Gillespie SE, Lecavalier L. Clinical and Demographic Correlates of Insomnia Symptoms in Children with Autism Spectrum Disorder. J Autism Dev Disord. 2025 Jul 31. doi: 10.1007/s10803-025-06944-3. Online ahead of print. No abstract available. PMID 40742672